CLINICAL TRIAL: NCT04827329
Title: Anesthetic Management of Patients With Chronic Sleep Disorders
Acronym: ANEST-SLEEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0192
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Narcolepsy; Idiopathic Hypersomnia; Restless Legs Syndrome
Keywords: Sleep; Anesthesia; Sedation; Surgery; drugs
MeSH Terms: conditions — Narcolepsy; Idiopathic Hypersomnia; Restless Legs Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a sleep disorder: Patients with a sleep disorder recording performed in the Sleep Unit in Montpellier University Hospital.
  Interventions: Other: Questionnaire
- Patients with a narcolepsy: Patients with a narcolepsy (type 1 or type 2) / a idiopathic hypersomnia or a restless legs syndrome.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will complete a questionnaire regarding their anesthesia history, course and possible complications, and Questions about their treatment for their sleep disorder.

SUMMARY:
The aim of this study is to describe and compare the anaesthesia history and possible problems encountered in 3 groups of patients with 3 chronic sleep diseases: narcolepsy, idiopathic hypersomnia, and restless legs syndrome followed at the Montpellier Sleep Unit.

For each participant, existing data from the medical record will be used, with their consent. All participants will complete a standardized questionnaire, concerning their history of anaesthesia, the course and possible complications, and questions about their treatment for their sleep disorder.

DETAILED DESCRIPTION:
This is both a retrospective and prospective single-center study. In the prospective part of the study, patients complete a self-questionnaire, with :

* a non-specific part, concerning the history of anaesthesia (locoregional or general), the patient's feelings about these anaesthesias (possible difficulties in waking up, pain) and details about the the course of the anaesthesia (including possible complications).
* a part specific to the sleep disease (possible rebound of symptoms, management of sleep treatments before and after anesthesia, sleep treatments before and after the different types of anesthesia).

Evaluation Criteria:

Main:

Frequency of history of locoregional and general anesthesia, and their possible complications.

Secondary:

Frequency of patients with rebound symptoms, or with worsening symptomatology (in each of the 3 groups, and in subgroups of patients with the same treatments), during locoregional and general anesthesia independently.

Other parameters collected via self-questionnaire (and at the time of the initial evaluation, retrospectively on medical records):

* Sociodemographic data: age, gender, body mass index
* Data related to the disease: age of onset of symptoms, age of diagnosis
* Other associated medical conditions
* Type of surgery
* Type, date and the number of anesthesia: locoregional, general

ELIGIBILITY:
Inclusion criteria:

* men and women, more than 16 years old
* diagnosed with a chronic sleep disorder including : Narcolepsy type 1, type 2, idiopathic hypersomnia, restless legs syndrome (diagnosis according to international criteria, ICSD-3, AASM, 2014).
* followed at Monpellier Sleep Disorders Unit.

Exclusion criteria:

- less than 16 years old at time of the study

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients, older than 16 years at time of the study, diagnosed with a sleep disorder: narcolepsy (1 or 2), idiopathic hypersomnia and restless legs syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency of history of locoregional | 1 day
  Frequency of history of locoregional and general anesthesia, and their possible complications : change in frequency or complication of symptoms after a surgical procedure under general or locoregional anesthesia

SECONDARY OUTCOMES:
Frequency of patients with rebound symptoms, or with worsening symptomatology | 1 day
  rebound of symptoms, occurrence of new symptoms or worsening of symptoms after a surgical procedure under general or locoregional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Hershner S, Kakkar R, Chung F, Singh M, Wong J, Auckley D. Narcolepsy, Anesthesia, and Sedation: A Survey of the Perioperative Experience of Patients With Narcolepsy. Anesth Analg. 2019 Nov;129(5):1374-1380. doi: 10.1213/ANE.0000000000003954. PMID 30540615
- [Result] Hershner S, Dauvilliers Y, Chung F, Singh M, Wong J, Gali B, Kakkar R, Mignot E, Thorpy M, Auckley D. Knowledge Gaps in the Perioperative Management of Adults With Narcolepsy: A Call for Further Research. Anesth Analg. 2019 Jul;129(1):204-211. doi: 10.1213/ANE.0000000000004088. PMID 30882519
- [Result] Ohshita N, Yamagata K, Himejima A, Kaneda K, Yasutome T, Matsuda Y, Tsutsumi YM, Momota Y. Anesthetic Management of a Patient With Restless Legs Syndrome: A Case Report. Anesth Prog. 2020 Dec 1;67(4):226-229. doi: 10.2344/anpr-67-02-10. PMID 33393604
- [Result] Raux M, Karroum EG, Arnulf I. Case scenario: anesthetic implications of restless legs syndrome. Anesthesiology. 2010 Jun;112(6):1511-7. doi: 10.1097/ALN.0b013e3181de2d66. No abstract available. PMID 20463578